CLINICAL TRIAL: NCT07022808
Title: Tele-Exercise to Promote Empowered Movement in Individuals With Spinal Cord Injury, TEEMS
Brief Title: Tele-Exercise to Promote Empowered Movement in Individuals With Spinal Cord Injury
Acronym: TEEMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Congressionally Directed Medical Research Progam (Unknown)
Responsible Party: Principal Investigator, Margaret A. Finley, Associate Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC40042_RCT_TEEMS; HT94252510367 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: randomized control trial; spinal cord injury; physical activity; tele-exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: A parallel group mixed methods randomized control trial comparing participation in the TEEMS program with exercise via asynchronous video library equivalent (control). The use of mixed methods will allow for the integration of quantitative findings with the qualitative, lived perspective of participants to provide a comprehensive analysis of the tele-exercise program outcomes.
Who Masked: Outcomes Assessor
Masking Description: biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Group Exercise (Experimental): All participants will participate in the TEEMS biweekly for 8 weeks (synchronous intervention or asynchronous video library). Participants will participate in the TEEMS biweekly for 8 weeks (synchronous intervention). The synchronous group will attend sessions 2 times per week, with all sessions recorded. The sessions will be 60-minutes total, including 45-minutes of physical activity. Recorded sessions will be made available for participants to use on their own at the end of each week, building a video of 16 videos. The program will be taught by a rehabilitation clinician with expertise in SCI and adapted exercise while our co-instructor will offer peer guidance and demonstrate lived translation of movement with an SCI. Class will take place over a web-based platform (such as Zoom).TEEMS instructors also orient participants to the Borg Rate of Perceived Exertion (RPE, 6-20 scale) to be used as an self-exertion check throughout class and to be recorded in a provided logbook. RPE is u
  Interventions: Other: Synchronous Group exercise
- Asynchronous Exercise (Active Comparator): The asynchronous control condition will be delivered using a private Youtube playlist. The asynchronous group will be provided with 2 recorded TEEMS videos weekly that align with the synchronous group sessions, building a 16 video library. Participants will participate in the TEEMS biweekly for 8 weeks (synchronous intervention). The asynchronous group will perform sessions 2 times per week. The sessions will be 60-minutes total, including 45-minutes of physical activity.
  Interventions: Other: Asynchronous exercise (Control)

INTERVENTIONS:
Other: Synchronous Group exercise — Participants will participate in the TEEMS biweekly for 8 weeks (synchronous intervention). The synchronous group will attend sessions 2 times per week, with all sessions recorded. The sessions will be 60-minutes total, including 45-minutes of physical activity. Recorded sessions will be made available for participants to use on their own at the end of each week, building a video of 16 videos. The program will be taught by a rehabilitation clinician with expertise in SCI and adapted exercise while our co-instructor will offer peer guidance and demonstrate lived translation of movement with an SCI. Class will take place over a web-based platform (such as Zoom).TEEMS instructors also orient participants to the Borg Rate of Perceived Exertion (RPE, 6-20 scale) to be used as an self-exertion check throughout class and to be recorded in a provided logbook. RPE is used as a self-assessment of moderate-vigorous intensity exercise.
  Arms: Synchronous Group Exercise
Other: Asynchronous exercise (Control) — Participants will participate in the TEEMS biweekly for 8 weeks (asynchronous video library). The asynchronous, control group will be provided with 2 recorded videos weekly that align with the synchronous group sessions, building a 16 video library as well. The sessions will be 60-minutes total, including 45-minutes of physical activity. The program will be taught by a rehabilitation clinician with expertise in SCI and adapted exercise while our co-instructor will offer peer guidance and demonstrate lived translation of movement with an SCI. Class will take place over a web-based platform (such as Zoom).TEEMS instructors also orient participants to the Borg Rate of Perceived Exertion (RPE, 6-20 scale) to be used as an self-exertion check throughout class and to be recorded in a provided logbook. RPE is used as a self-assessment of moderate-vigorous intensity exercise.
  Arms: Asynchronous Exercise

SUMMARY:
To achieve our specific aims and hypotheses we will conduct a parallel group mixed methods randomized control trial comparing participation in the TEEMS program with exercise via asynchronous video library equivalent (control). The use of mixed methods will allow for the integration of quantitative findings with the qualitative, lived perspective of participants to provide a comprehensive analysis of the tele-exercise program outcomes. All aspects of the study from recruitment, screening, data collection, tele-exercise delivery and team meetings will be virtual to promote access and inclusion by removing barriers and promoting engagement. This study will compare our live group TEEMS program with individual pre-recorded exercise videos. We created TEEMS with the intention of maximizing exercise independence for participants, which decreases need for caregivers during physical activity. The design and participation in TEEMS is meant to increase personal factors that facilitate participation in exercise. These personal factors include confidence and positive associations with exercise. When these personal factors are targeted, individuals with SCI are more likely to participate in physical activity, which supports overall health and QoL.

DETAILED DESCRIPTION:
Background: Over half of individuals with spinal cord injury (SCI) report no regular physical activity, a cornerstone for independent function and psychosocial health. Studies confirm comparable prevalence and disruptive impact of SCI inactivity/sedentary lifestyle in the civilian and military community, as well as similar barriers to exercise participation. The proposed study will simultaneously address barriers and promote facilitators of physical activity behavior through expert SCI-specific knowledge, peer mentoring, group cohesion, creating autonomy and self-efficacy, mechanisms of engagement that are relevant across both military and civilian sectors.

Hypothesis/Objectives: Our broad research objective is to determine the effectiveness of a novel group exercise program, (Tele Exercise to promote Empowered Movement with Spinal Cord Injury, TEEMS) that will foster the development of lifelong physical activity behavior by enhancing self-efficacy, specifically as it pertains to exercise. This is facilitated through expert knowledge translation with peer interaction and mentoring. We hypothesize that greater improvements in physical activity participation and psychosocial determinants will be found following participation in TEEMS compared to the control group and will be retained at 16-weeks.

Specific Aims: Aim 1-3 will determine if participation in the synchronous TEEMS program improves psychosocial determinants (self-efficacy, outcome expectations, resilience, kinesiophobia, quality of life) of physical activity behavior (weekly minutes by self-report, wearable activity monitor) and physical factors (pain behaviors, mobility and sleep disturbance) compared to an asynchronous video program (control). Narrative accounts will elaborate on quantitative findings of psychosocial impact of TEEMS participation. Aim 4 will integrate quantitative findings with qualitative, narrative themes of participation in TEEMS to allow for a comprehensive understanding of the impact of group tele-exercise participation compared to an asynchronous video program.

Study Design: We will conduct a randomized control trial using a parallel mixed methods design comparing synchronous participation in the TEEMS program with exercise via asynchronous videos (control). Per the mixed methods design the two distinct datasets (quantitative and qualitative) will be independently collected and analyzed in parallel, with the goal of convergent integration. Data will be collected pre-program, post-program (8-weeks) at retention at 16-weeks. Our novel remotely delivered, synchronous tele-exercise program reduces barriers to access and provides peer support in an inclusive SCI-specific program led by experts in adapted exercise and co-led by individuals living with SCI. Our program conceptual framework is Social Cognitive Theory (SCT), which emphasizes that influencing sociostructural factors and personal determinants will impact health behaviors including physical activity. Each class will be recorded and upon request, participants will be provided access if they choose to perform a class independently. The control group will receive a bank of 16 videos from the previous 8-week session of the tele-exercise program, with a goal of completing 2 videos/week. They will be provided with instructions on progression through the videos and as with the intervention group access as well as ability to access if they choose to perform a class independently. The control group will have weekly communication with the investigative team as well as one-on-one sessions with the leader and co-leader at baseline, week 3 and week 6 to discuss progression and received feedback. All research activities (recruitment, enrollment, communication, data collection, intervention) will be conducted remotely through web-enhanced video systems (Zoom).

ELIGIBILITY:
Inclusion Criteria:

1. at least 12 months post SCI (motor spinal level C5 or below)
2. between 18-75 years of age
3. ability to elevate shoulders >25% range
4. use assistive technology for mobility
5. not currently receiving structured rehabilitation (i.e. new episode of inpatient or outpatient rehabilitation services to treat a new or exacerbated mobility issue. Individuals attending outpatient services for ongoing wellness reasons are eligible to participate).
6. screened and medically cleared (if appropriate) for participation using the American College of Sports Medicine (ACSM) Preparticipation Health Screening Tool. The ACSM Health Screen helps to determine if an individuals should seek a medical referral prior to participation in exercise. The guideline for the screening are based on (1) current exercise participation, (2) history and symptoms of cardiovascular, metabolic, or renal disease, and (3) desired exercise intensity. The algorithm is based on risk stratification and minimizing the barriers of exercise participation by decreasing the number of unnecessary medical referrals.

   For this study and the safety of participants, those who need a medical referral based on the ACSM preparticipation health screen will be required to provide documentation of medical clearance from their primary medical provider prior to study participation. Dr. York will review screening information and medical clearances to ensure safe inclusion.
7. internet access to attend synchronous exercise classes

Exclusion Criteria:

1. Known or suggestive cardiovascular, metabolic, and/or renal disease and/or presence of absolute or relative contraindications to exercise participation that is considered unsafe by their medical team
2. self-report previous hospitalization within a month,
3. self report active pressure injury
4. self report recent osteoporotic fracture
5. self-report uncorrectable vision loss,
6. self-report preexisting neurological conditions other than SCI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Exercise Self Efficacy | at baseline (enrollment), 8-weeks, 16-weeks
  The SCI Exercise Self-efficacy Scale (ESES).This self-report measures the construct of self-efficacy, or personal beliefs in one's capabilities relating to exercise participation in individuals with SCI. Self-efficacy is cited as the most critical personal factor to behavior change. This outcome demonstrates reliability and high internal consistency.
Exercise Outcome Expectations | baseline (enrollment), 8-weeks and 16-weeks
  The Multidimensional Outcome Expectations for Exercise Scale (MOEES). This self-report measure addresses physical, social, and self-evaluative components of outcome expectations, another critical element needed for health behavior change. This tool also demonstrates high internal consistency and validity
Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) | baseline (enrollment), one -week, 8-weeks, 16-weeks
  The Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) is an SCI-specific, self-report measure of leisure-time physical activity that assesses minutes of mild, moderate, and heavy intensity leisure-time physical activity performed over the previous 7-days. Test-retest reliability and criterion validity of the LTPAQ-SCI has been established. The LTPAQ will be obtained an additional time following participation in the first tele-exercise class.
Physical Activity Measure. | baseline (enrollment), 8-weeks, 16-weeks
  Physical Activity monitoring: To assess physical activity engagement, mobility function monitoring will be performed by using an activity monitor (GENEActiv) placed on the non-dominant wrist of the individual over a duration of 7 days (matching the duration of the self-report LTPAQ).
Subjective Quality of Life Questionnaire (SQoL) | baseline (enrollment), 8-weeks, 16-weeks
  This questionnaire is a global measure of subjective perception of QoL. The scale is a Likert-type scale measuring satisfaction with life as a whole: Participants are asked to take everything in their life into account and rate it on an ordinal scale from 1 (life is very distressing; it's hard to imagine how it could get much worse) to 7 (life is great; it's hard to imagine how it could get much better).
Qualitative data | baseline, 8-weeks
  Focus group data collection will be conducted via secure web-based video conferencing platform (Zoom). Data will be obtained at pre-program and post-program (8-weeks). All participants will join focus group interviews of 5-8 individuals that will take approximately 60 minutes pre (baseline) and post- program (8-weeks). Focus groups will be facilitated by a trained team member and co- facilitated by a lived experience class co-instructor . The open-ended guiding questions will be grounded by the numeric outcomes corresponding to measurement constructs and our previous work.

SECONDARY OUTCOMES:
Loneliness (UCLA Loneliness Scale) - | baseline (enrollment), 8-weeks
  Loneliness (UCLA Loneliness Scale) - This 20-item measure assesses constructs of loneliness including interpersonal relationships, health, and wellbeing.
Pain phenomena (SCIQOL-PP) | baseline (enrollment), 8-weeks
  Pain interference and Pain Behavior10 Within the ICF domains of activity and participation, the SCI-QOL measurement system is comprised of 19 item response theory (IRT) calibrated banks/scales across physical, emotional, and social functioning. Each bank is available in a short form (7-10 questions). In clinical or research context, the SCI-QOL is used to document the initial impact of SCI, changes and trajectories. The SCIQOL pain phenomena (pain behavior and pain interference) representing the domain of physical health will be a primary measure. SCIQOL Pain Interference short form (10 items) and the SCIQOL Pain Behavior scale (7 items) are versions of the PROMIS Pain Interference and Pain Behavior item banks, respectively, that have been optimized for individuals with SCI.
Self-esteem (SCI-QOL-SE) | baseline (enrollment), 8-weeks
  Self-esteem (SCI-QOL-SE)- The Self-Esteem bank of 8 items assesses emotional, evaluative, and cognitive perceptions of personal competence and worth. This self-evaluation provides a reference by which to compare oneself to relevant others in social and socially competitive situations
Depression (SCI-QOL-DEPR) | baseline (enrollment), 8-weeks
  Depression (SCI-QOL-DEPR)6-This 10-item short form contains items addressing despair and/or a loss of interest in things as well as feelings of hopelessness, helplessness, and worthlessness the individual has experienced in the past 7 days.
Resilience (SCI-QOL-RES) | baseline (enrollment), 8-weeks
  Resilience (SCI-QOL-RES)- The Resilience short form bank contains 8 items that address issues such as motivation, coping, and acceptance.
Participation in Social Roles and Activity (SCI-QOL-PSR) | baseline (enrollment), 8-weeks
  Participation in Social Roles and Activity (SCI-QOL-PSR) - This domain describes the degree of current involvement in social roles, activities, and responsibilities, including work, family, friends and leisure over the past 7 days in a 10-item question bank
Satisfaction with Social Roles and Activity (SCI-QOL-SSR) | baseline (enrollment), 8-weeks
  Satisfaction with Social Roles and Activity (SCI-QOL-SSR)- The satisfaction with social roles and activity short form contains 10 items with reference to the individual's satisfaction and disappointment with involvement in usual social roles, activities, and responsibilities, including work, family, friends and leisure in the past 7 days.
General Sleep Disturbance Scale | baseline (enrollment), 8-weeks
  General Sleep Disturbance Scale: The GSDS is a 21-item scale was designed to evaluate the incidence and nature of sleep disturbances. Questions pertain to a variety of general sleep issues, including problems initiating sleep, waking up during sleep, waking too early from sleep, quality of sleep, quantity of sleep, fatigue and alertness at work, and the use of substances to induce sleep. The GSDS queries respondents regarding the frequency with which they've experienced certain sleep difficulties within the previous week. Respondents use an eight-point, Likert-type scale ranging from 0 (meaning "never") to 7 ("every day") to respond to each item.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Finley, PT, PhD, Principal Investigator — Drexel University; Laura Baehr, PT, DPT, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University Health Science Building, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the FAIR practices and standards for sharing of SCI data, we will share final de-identified individual participant outcomes and metadata organized as recommended by ODC-SCI, using formatting standards established by the ODC-SCI. By following these recommendations, we will ensure that our data may be harmonized with other clinical studies and has passed community quality checks. All experimental data will be accompanied by a detailed experimental protocol and additional data and metadata. The protocols will be linked to the experimental data both in the publication and the data sharing platform. ODC-SCI requires the publication of a data dictionary that defines all variables present in the data set in a standard format.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of the research, quantitative data will be made available through the Open Data Commons for Spinal Cord Injury (ODC-SCI). We will make our data available on the public site upon submission of a pre-print or publication of the study in a peer-reviewed journal. ODC-SCI fully supports peer review by providing a private space which can be accessed anonymously by peer reviewer issued provisional DOIs. These can be used to hold the data under embargo before release. If the study is not successful and/or we do not publish the study, we will still make our negative data available through ODC-SCI.
Access Criteria: We will make our data available through ODC-SCI under an open CC-BY license. The ODC-SCI is compliant with requirements for FAIR and trustworthy repositories established by NIH, NLM and journals. ODC-SCI runs an open-source cloud- based platform optimized for managing and sharing multimodal data